CLINICAL TRIAL: NCT02378844
Title: A Randomized, Multicentre, Double-blind, Parallel, Sham-controlled Study of gammaCore®, a Non-invasive Vagal Nerve Stimulator (nVNS), for Prevention of Episodic Migraine
Brief Title: A Randomized, Sham-controlled Study of gammaCore ® (nVNS) for Prevention of Episodic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GM-11
Record Dates: First submitted 2015-02-18; First posted 2015-03-04 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gammaCore®-R (Active Comparator): Subjects will be instructed to treat three times per day, 2 consecutive bilateral stimulations, upon waking, six to eight hours following the first daily treatment, and six to eight hours following the second daily treatment (one stimulation on the right side immediately followed by a second stimulation on the left side).
  Interventions: Device: gammaCore®-R
- gammaCore®-R Sham (Sham Comparator): Subjects will be instructed to treat three times per day, 2 consecutive bilateral stimulations, upon waking, six to eight hours following the first daily treatment, and six to eight hours following the second daily treatment (one stimulation on the right side immediately followed by a second stimulation on the left side).
  Interventions: Device: gammaCore®-R Sham

INTERVENTIONS:
Device: gammaCore®-R — Subjects will be instructed to treat three times per day, 2 consecutive bilateral stimulations, upon waking, six to eight hours following the first daily treatment, and six to eight hours following the second daily treatment (one stimulation on the right side immediately followed by a second stimulation on the left side).
  Arms: gammaCore®-R
Device: gammaCore®-R Sham — Subjects will be instructed to treat three times per day, 2 consecutive bilateral stimulations, upon waking, six to eight hours following the first daily treatment, and six to eight hours following the second daily treatment (one stimulation on the right side immediately followed by a second stimulation on the left side).
  Arms: gammaCore®-R Sham

SUMMARY:
A prospective, double-blind, randomized, sham-controlled, multicentre investigation.

DETAILED DESCRIPTION:
The study period will begin with a four week run-in period, during which there is no investigational treatment. The purpose of the run-in period will be observation for baseline comparison.

The run-in period will be, followed by a 12 week randomized period when the subjects will be randomized (1:1) to either active treatment or sham (inactive) treatment.

The randomized period will be followed by a 24 week open label period, where the subjects in the sham treatment group will switch in treatment assignment and receive a gammaCore®-R and the gammaCore®-R will continue to receive an active treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Is between the ages of 18 and 75 years.
2. Has been previously diagnosed with migraine (with or without aura) in accordance with the International Classification of Headache Disorders (ICHD)-3 Beta Classification criteria.
3. Experience between 5 and 12 migraine days per month (over the last 4 months) with at least 2 of the migraines lasting more than 4 hours.
4. Has age of onset of migraine less than 50 years old.
5. Agrees not to use any migraine prevention treatments (including Botox injections) and/or medications (exclusive of medications taken for acute relief of migraine symptoms).
6. Agrees to refrain from initiating or changing the type, dosage or frequency of any prophylactic medications for indications other than migraine that in the opinion of the clinician may interfere with the study objectives (e.g. antidepressant, anti convulsant, beta blockers, etc.).
7. Agrees to use the gammaCore®-R device as intended, follow all of the requirements of the study including follow-up visit requirements, record required study data in the subject dairy, and other self-assessment questionnaires.
8. Is able to provide written Informed Consent.

Exclusion Criteria:

1. Has a concomitant medical condition that will require oral or injectable steroids during the study.
2. Has a history of any intracranial aneurysm, intracranial haemorrhage, brain tumour or significant head trauma.
3. Has a structural abnormality at the gammaCore®-R treatment site (e.g lymphadenopathy previous surgery or abnormal anatomy).
4. Has pain at the gammaCore®-R treatment site (e.g.dysesthesia, neuralgia and/or cervicalgia).
5. Has other significant pain problem (e.g.cancer pain, fibromyalgia or other head or facial disorder) that in the opinion of the investigator may confound the study assessments
6. Has know or suspected severe cardiac disease(e.g. symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure (CHF)).
7. Has known or suspected severe cerebrovascular disease, (e.g. prior stroke or transient ischemic attack, symptomatic carotid artery disease, prior carotid endarterectomy or other vascular neck surgery).
8. Has an abnormal baseline Electrocardiogram (ECG) e.g. second and third degree heart block, prolonged QT interval, atrial fibrillation, atrial flutter, history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction).
9. Has had a cervical vagotomy.
10. Has uncontrolled high blood pressure (systolic >160 diastolic > 100 after 3 repeated measurements within 24 hours).
11. Is currently implanted with an electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator cochlear implant, Sphenopalatine ganglion stimulator or Occipital nerve stimulator).
12. Has been implanted with metal cervical spine hardware or has a metallic implant near the gammaCore®-R stimulation site.
13. Has a known history of suspicion of secondary headache.
14. Has a history of syncope (within the last five years).
15. Has a history of seizures (within the last five years).
16. Has a known or suspicion of substance abuse or addiction (within the last 5 years).
17. Is using marijuana (including medical marijuana) for any indications, more than twice a month.
18. Currently takes simple analgesics or non-steroidal anti-inflammatory drugs (NSAIDs) greater than 15 days per month or triptans, ergots or combined analgesics greater than 10 days per month for headaches or other body pain.
19. Currently takes prescription opioids greater than 2 days per month for headaches or body pain.
20. Has taken medications for migraine prophylaxis in the previous 30 days.
21. Has previous diagnosis of medication overuse headache (MoH) , which has reverted to episodic migraine within the last 6 months.
22. Meets the ICHD-3 Beta Classification criteria for chronic migraine (> 15 headache days per month).
23. Has failed an adequate trial (two months or greater) of at least 3 classes of a drug therapy for the prophylaxis of migraine .
24. Has had surgery for migraine prevention.
25. Has undergone nerve block (occipital or other) in the head or neck within the last 2 months.
26. Has received Botox injections within the last 6 months.
27. Is pregnant or thinking of becoming pregnant during the study period, or of childbearing years and is unwilling to use and accepted form of birth control.
28. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
29. Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self- assessments is compromised (e.g. homeless, developmentally disabled and prisoner).
30. Is a relative of or an employee of the investigator or the clinical study site.
31. Has psychiatric or cognitive disorder and/or behavioural problems which in the opinion of the clinician may interfere with the study.
32. Has previously used the gammaCore® device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Diener, Professor, Principal Investigator — Universtätsklinikum Essen
Locations (22):
- Neurology Department, University of Liège, Liège, Belgium
- Danish Headache Center, Glostrup Municipality, Denmark
- Germany (7):
  - Neurologische Klinik und Poliklinik, Charité Campus Mitte, Berlin
  - Klinik für Neurologie, Universitätsklinikum Essen, Essen
  - CTC, University Medical Center Hamburg-Eppendorf, Hamburg
  - Migräne- und Kopfschmertzklinik Königstein, Königstein
  - Klinik für Neurologie, Ludwig-Maximilliams-Universität, Klinikum Grosshadern, München
  - Zentrum für Neurologie und Epileptologie, Hertie-Institut für Klinische Hirnforschung, Tübingen
  - DKD HELIOS Klinik Wiesbaden, Wiesbaden
- Neurology Department, Athens Naval Hospital, Athens, Greece
- Neurology Department, Leiden University Center, Leiden, Netherlands
- Sandvika Nevrosenter AS, Sandvika, Norway
- Spain (4):
  - Headache Unit, University Hospital Vall d'Hebron, Barcelona
  - Servicio de Neurologia, Hospital Ruber Internacional, Madrid
  - Servicio de Neurologia, Clinica Universidad de Navarra, Pamplona
  - Servicio de Neurologia, Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (6):
  - Basildon University Hospital, Basildon, Essex
  - School of Clinical and Expermental Medicine, Birmingham
  - Neurology Department, The Southern Hospital, Glasgow
  - Neurology Department, Hull Royal Infirmary, Hull
  - Neurology Department, The Walton Center, Liverpool
  - Neurology Department, King's College London, London

IPD SHARING:
Plan to Share IPD: No
Results from the whole study will published but not individual participant data.

REFERENCES:
- [Derived] Diener HC, Goadsby PJ, Ashina M, Al-Karagholi MA, Sinclair A, Mitsikostas D, Magis D, Pozo-Rosich P, Irimia Sieira P, Lainez MJ, Gaul C, Silver N, Hoffmann J, Marin J, Liebler E, Ferrari MD. Non-invasive vagus nerve stimulation (nVNS) for the preventive treatment of episodic migraine: The multicentre, double-blind, randomised, sham-controlled PREMIUM trial. Cephalalgia. 2019 Oct;39(12):1475-1487. doi: 10.1177/0333102419876920. Epub 2019 Sep 15. PMID 31522546

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Randomized: Subjects that were screen failures and were not randomized
Period: Run-in Period
Arm/Group | gammaCore®-R | gammaCore®-R Sham | Not Randomized
Started | 169 | 172 | 136
Completed | 165 | 167 | 0
Not Completed | 4 | 5 | 136
Period: Randomized Period (Double Blind)
Arm/Group | gammaCore®-R | gammaCore®-R Sham | Not Randomized
Started | 165 | 167 | 0
Completed | 142 | 135 | 0
Not Completed | 23 | 32 | 0
Period: Open Label Period
Arm/Group | gammaCore®-R | gammaCore®-R Sham | Not Randomized
Started | 142 | 135 | 0
Completed | 99 | 87 | 0
Not Completed | 43 | 48 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population, Intention to Treat (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | gammaCore®-R | gammaCore®-R Sham | Total
Number analyzed (Participants) | 165 | 167 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] — Year of inclusion minus date of birth
  years | 43.5 (11.11) | 41.4 (12.26) | 42.4 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex, male or female, reported at time of inclusion in study
  Participants
    Female | 142 | 138 | 280
    Male | 23 | 29 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity recorded at time of inclusion into study
  Participants
    Race: Caucasian | 160 | 154 | 314
    Race: Black | 0 | 2 | 2
    Race: Asian | 1 | 3 | 4
    Race: Other | 4 | 8 | 12
Region of Enrollment [Number; unit: participants] — Numbers of enrolled subjects per country
  participants
    Greece | 15 | 16 | 31
    Netherlands | 15 | 16 | 31
    Belgium | 11 | 11 | 22
    Norway | 6 | 6 | 12
    Denmark | 17 | 16 | 33
    United Kingdom | 43 | 48 | 91
    Germany | 36 | 32 | 68
    Spain | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Migraine Days
Description: Change in number of migraine days (as reported in subject diary), comparing the 4 week run-in period to the last 4 weeks in the randomized period.
Time Frame: last 4 weeks of the randomized/controlled period compared to the subject's own 4-week run-in period.
Population: Randomized population, Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | gammaCore®-R | gammaCore®-R Sham
Number analyzed (Participants) | 165 | 167
Days | -1.98 (3.031) | -1.53 (3.090)

2. Secondary Outcome: Number of Participants With 50% Responder Rate
Description: The number of subjects with a reduction of 50% or more in number of migraine days (as reported in the subject diary) from the run-in period to the last 4 weeks of the double-blind period.
Time Frame: The last four weeks in the randomization period compared to the four week run-in period.
Population: Randomized population, Intention to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore®-R | gammaCore®-R Sham
Number analyzed (Participants) | 165 | 167
Participants | 47 | 38

3. Secondary Outcome: Mean Change in Number of Headache Days
Description: The mean change in number of headache days (as reported in the subject diary) from the run-in period to the last 4 weeks of the double-blind period.
Time Frame: The last four weeks in the randomization period compared to the four week run-in period.
Population: Randomized population, Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | gammaCore®-R | gammaCore®-R Sham
Number analyzed (Participants) | 165 | 167
Days | -2.28 (3.623) | -1.72 (3.732)

4. Secondary Outcome: Change in Number of Acute Medication Days
Description: The mean change in number of acute medication days (as reported in the subject diary) from the run-in period to the last 4 weeks of the double-blind period
Time Frame: The last four weeks in the randomization period compared to the four week run-in period.
Population: Randomized population, Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: acute medication days
Arm/Group | gammaCore®-R | gammaCore®-R Sham
Number analyzed (Participants) | 165 | 167
acute medication days | -1.65 (3.310) | -1.02 (3.310)

5. Secondary Outcome: Change in Headache Disability Using Headache Impact Test-6
Description: Change in headache disability from the 4 week run-in period to the last 4 weeks of the randomized period as measured using the Headache Impact Test-6 (HIT-6). The HIT-6 measures the impact if a subject's headaches on their ability to function at work, at home and in social situations. Subjects are presented with 6 questions about ability to function and normal daily life and for each question they rate the impact of their headaches as 'never' (6 points) or 'rarely' (9 points) or 'sometimes' (10 points) or 'very often' (11 points) or 'always' (13 points). Minimum score = 36, maximum score = 78. A higher score indicates more impact.
Time Frame: From four week run-in period to last four weeks in the randomization period
Population: Randomized population, Intention to Treat (ITT) In the active group 23 subjects had missing data, in the sham group 32 subjects had missing data at the end of the randomized period
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | gammaCore®-R | gammaCore®-R Sham
Number analyzed (Participants) | 165 | 167
units on a scale
  HIT-6 score Run-in perio | 63.442 [49 to 74] | 64.263 [44 to 76]
  HIT-6 score end of Randomized period: number analyzed (Participants) | 142 | 135
  HIT-6 score end of Randomized period | 60.234 [42 to 76] | 60.992 [40 to 78]

6. Secondary Outcome: Number of Participants According to Grade on the Migraine Disability Assessment (MIDAS) Before and After Randomized Period
Description: Migraine Disability Assessment (MIDAS) score from the end of run-in period to the end of randomized period. The MIDAS assessment measures the effect of headaches on a subject's daily functioning. It takes into account the past 3 months and is comprised of five questions. A lower score indicated less disability, a higher score indicates more disability. The scores are graded:
  0-5, MIDAS Grade I, little disability 6-10, MIDAS Grade II, mild disability 11 to 20 MIDAS Grade III, moderate disability 21+ MIDAS Grade IV, severe disability
Time Frame: 3 months - end of run-in period to end of randomized period
Population: Randomized population, Intention to Treat (ITT) At randomisation (visit 2) subject numbers are 165 gammaCore-R and 167 gammaCore-R Sham.
  At visit 6 the numbers are lower due to early subject discontinuation: 141 gammaCore-R and 132 gammaCore-R Sham
Measure: Number; unit: participants
Arm/Group | gammaCore®-R | gammaCore®-R Sham
Number analyzed (Participants) | 165 | 167
participants
  Week 0 of Randomized Period (Visit 2) Grade I | 11 | 11
  Week 0 of Randomized Period (Visit 2) Grade II | 15 | 15
  Week 0 of Randomized Period (Visit 2) Grade III | 23 | 32
  Week 0 of Randomized Period (Visit 2) Grade IV | 116 | 109
  Week 12 (Visit 6) Grade I: number analyzed (Participants) | 141 | 132
  Week 12 (Visit 6) Grade I | 22 | 24
  Week 12 (Visit 6) Grade II: number analyzed (Participants) | 141 | 132
  Week 12 (Visit 6) Grade II | 19 | 17
  Week 12 (Visit 6) Grade III: number analyzed (Participants) | 141 | 132
  Week 12 (Visit 6) Grade III | 37 | 27
  Week 12 (Visit 6) Grade IV: number analyzed (Participants) | 141 | 132
  Week 12 (Visit 6) Grade IV | 63 | 64

7. Secondary Outcome: Compare Changes in Quality of Life EuroQol Questionnaire 5 Dimensions and 5 Levels (EQ-5D-5L)
Description: The descriptive system comprises five dimensions (5D): mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension has 5 levels (5L): no problems (1) , slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5).
  Minimum score is 5 (no problems) and maximum score is 25 (extreme problems)
  An overall health question is asked using a visual analogue scale(VAS) from 0-100 where 0 is bad health and 100 good health
Time Frame: From four week run-in period to last four weeks in the randomization period
Population: Randomized population, Intention to Treat (ITT) In the active group 24 subjects had missing data, in the sham group 35 subjects had missing data at the end of the randomized period
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | gammaCore®-R | gammaCore®-R Sham
Number analyzed (Participants) | 165 | 167
scores on a scale
  Mobility run-in period | 1.10 [1 to 4] | 1.10 [1 to 3]
  Mobility randomized period: number analyzed (Participants) | 141 | 132
  Mobility randomized period | 1.09 [1 to 3] | 1.07 [1 to 3]
  Selfcare run-in period | 1.02 [1 to 4] | 1 [1 to 1]
  Selfcare randomized period: number analyzed (Participants) | 141 | 132
  Selfcare randomized period | 1.02 [1 to 3] | 1.02 [1 to 3]
  Usual activities run-in period | 1.27 [1 to 5] | 1.23 [1 to 4]
  Usual activities randomized period: number analyzed (Participants) | 141 | 132
  Usual activities randomized period | 1.24 [1 to 3] | 1.22 [1 to 3]
  Pain/discomfort run-in period | 1.56 [1 to 5] | 1.59 [1 to 5]
  Pain/discomfort randomized period: number analyzed (Participants) | 141 | 132
  Pain/discomfort randomized period | 1.50 [1 to 4] | 1.48 [1 to 4]
  Anxiety/depression run-in period | 1.35 [1 to 4] | 1.4 [1 to 5]
  Anxiety/depression randomized period: number analyzed (Participants) | 141 | 132
  Anxiety/depression randomized period | 1.32 [1 to 3] | 1.41 [1 to 5]
  Visual analogue scale )VAS) run-in period | 80.97 [5 to 100] | 80.3 [8 to 100]
  Visual analogue scale (VAS) randomized period: number analyzed (Participants) | 141 | 132
  Visual analogue scale (VAS) randomized period | 82.46 [38 to 100] | 76.35 [30 to 100]

8. Secondary Outcome: Change in Migraine Days in the Open Label Period (Adjusted ANCOVA)
Description: Change in number of migraine days (as reported in subject diary) during the 6 month open label period compared to the baseline run-in period.
Time Frame: The 6 month open-label period compared to the four week run-in period
Population: Randomized population (Intent to treat)
Measure: Mean (Full Range); unit: Days
Arm/Group | gammaCore®-R | gammaCore®-R Sham
Number analyzed (Participants) | 165 | 167
Days
  Migraine days run in period | 7.94 [3 to 15] | 7.9 [3 to 12.9]
  Migraine days open label period | 5.75 [0 to 20] | 5.7 [0 to 17]

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse Effects were collected for all subjects for the duration of the study.
Time Frame: up to Week 36
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Open Label: Subjects will be instructed to treat three times per day, 2 consecutive bilateral stimulations, upon waking, six to eight hours following the first daily treatment, and six to eight hours following the second daily treatment (one stimulation on the right side immediately followed by a second stimulation on the left side).
Arm/Group | gammaCore®-R | gammaCore®-R Sham | Not Randomized | Open Label
Number analyzed (Participants) | 169 | 172 | 136 | 277
Participants
  Serious adverse events | 2 | 1 | 0 | 2
  Adverse events (non-serious) | 74 | 91 | 13 | 118

10. Secondary Outcome: Change in Headache Days in the Open Label Period
Description: The mean change in number of headache days (as reported in the subject diary) during the open label period compared to the base-line run-in period
Time Frame: The 6 month open-label period compared to the four week run-in period
Population: Randomized population (Intent to treat)
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | gammaCore®-R | gammaCore®-R Sham
Number analyzed (Participants) | 165 | 167
Days | -0.55 [-1.08 to -0.02] | -0.51 [-1.02 to -0.00]

ADVERSE EVENTS:
Time Frame: 40 weeks (run-in 4 weeks, double blind/randomized 12 weeks, open label 24 weeks)
Groups:
- Not Randomised: Subjects that were screen failures and were not randomized.
Arm/Group | gammaCore®-R | gammaCore®-R Sham | Not Randomised | Open Label
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/172 | 0/136 | 0/277
Serious Adverse Events (participants affected / at risk) | 2/169 | 1/172 | 0/136 | 2/277
Other Adverse Events (participants affected / at risk) | 74/169 | 91/172 | 13/136 | 118/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gammaCore®-R (N=169) | gammaCore®-R Sham (N=172) | Not Randomised (N=136) | Open Label (N=277)
Admitted because of suspecion of appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal Cell Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgery for removal cyste and twisted fallopian tube left (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
carrier BRCA2 gene, prophylactic surgery: adnex extirpation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
obstructive syndrom with dyspnea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gammaCore®-R (N=169) | gammaCore®-R Sham (N=172) | Not Randomised (N=136) | Open Label (N=277)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Adrenomegaly (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Conjunctival irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema eyelids (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (5)
Application site dermatitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site discolouration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site discomfort (General disorders) | 6 (6) | 3 (3) | 0 (0) | 2 (2)
Application site eczema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 3 (4) | 7 (9) | 0 (0) | 0 (0)
Application site injury (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 4 (4) | 8 (9) | 0 (0) | 0 (0)
Application site pain (General disorders) | 4 (4) | 7 (12) | 0 (0) | 4 (4)
Application site pruritus (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Application site rash (General disorders) | 1 (1) | 13 (14) | 0 (0) | 0 (0)
Application site reaction (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Application site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site pustules (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 11 (12) | 8 (8) | 0 (0) | 10 (13)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 22 (22) | 10 (10) | 3 (3) | 18 (21)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Q fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 4 (5)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Heart rate irregular (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 1 (1) | 4 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (10) | 3 (5) | 1 (1) | 6 (9)
Dysgeusia (Nervous system disorders) | 1 (1) | 8 (9) | 0 (0) | 2 (2)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 3 (3) | 4 (5) | 0 (0) | 3 (3)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Phantom pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Status migrainosus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Bruxism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphemia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6) | 0 (0) | 5 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne cystic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
Cyst removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oophorectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papilloma excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Preventive surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Labile blood pressure (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02378844/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT02378844/SAP_001.pdf